CLINICAL TRIAL: NCT00268242
Title: A Phase II Study of Gemcitabine/ Mitoxantrone in Patients With Acute Myeloid Leukemia in First Relapse
Brief Title: Gemcitabine and Mitoxantrone in Treating Patients With Relapsed Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: If </= 5 of the initial 18 patients had a CR, the study would be stopped. Only 5 patients (21%) of 24 enrolled patients had a CR so the study was terminated.
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE-CCF-7725; P30CA043703 (NIH); CASE-CCF-7725 (Other: Cleveland Clinic)
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2015-08

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7)
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Gemcitabine; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine + Mitoxantrone (Experimental): Gemcitabine Hydrochloride as administered as a continuous intravenous infusion (I.V.) at 10mg/m^2/minute for 12 hours, starting on Day 1. Mitoxantrone Hydrochloride was given at a dose of 12mg/m^2/day I.V. on days 1, 2, and 3.
  Interventions: Drug: Gemcitabine Hydrochloride; Drug: Mitoxantrone Hydrochloride

INTERVENTIONS:
Drug: Gemcitabine Hydrochloride — 10 mg/m2/ min IV for 12 hours
  Other Names: Gemcitabine
Drug: Mitoxantrone Hydrochloride — 12 mg/m2/day IV (administer over 30-60 minutes) on Day 1, 2 and 3
  Other Names: Mitoxantrone

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and mitoxantrone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with mitoxantrone works in treating patients with relapsed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete response (CR) rate (CR and incomplete blood count recovery (CRi)) of patients with acute myeloid leukemia in first relapse treated with gemcitabine hydrochloride and mitoxantrone hydrochloride.

Secondary

* Evaluate disease free and overall survival of patients with acute myeloid leukemia in first relapse treated with this particular chemotherapy regimen.
* Assess hematologic and non-hematologic toxicity associated with this regimen.
* Assess laboratory correlates of drug resistance in patients with relapsed acute myeloid leukemia.
* Assess the percentage of patients receiving subsequent bone marrow transplantation.

OUTLINE: This is an open-label, multicenter study.

Patients receive gemcitabine hydrochloride IV over 12 hours on day 1 and mitoxantrone hydrochloride IV over 30-60 minutes on days 1, 2, and 3. After completion of a single course of therapy, patients who achieve a complete response may receive 1 additional course of therapy at the discretion of the treating physician.

After completion of study treatment, patients are followed periodically for survival.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Bone marrow examination or peripheral blood analysis confirming active acute myeloid leukemia by WHO criteria

  * No M3 acute myeloid leukemia
* Not a candidate for allogenic bone marrow transplantation
* Patient must be in first relapse after having received induction chemotherapy

  * Received 1 or 2 courses with remission lasting at least 1 month
* Patients with chloromas or leukemia cutis are eligible
* No evidence of leptomeningeal involvement

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Liver enzymes (total bilirubin, aspartate aminotransferase (AST) and ALT) ≤ 2.5 times the upper limits of normal

  * Liver enzymes ≥ 2.5 are acceptable if physician documents that it is secondary to the disease
* Serum creatinine ≤ 3 mg/dL
* No poorly controlled medical conditions that would seriously complicate compliance with this study
* No other active primary malignancy other than carcinoma in situ of the cervix or basal cell carcinoma of the skin
* No New York Heart Association grade III or IV cardiac problems, defined as congestive heart failure or myocardial infarction within 6 months prior to start of study
* Pregnant or nursing women are ineligible
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No documented history of human immunodeficiency virus (HIV) infection
* No history of chronic liver disease
* Ejection fraction ≥ 45%
* No significant history of non-compliance to medical regimens or inability to give reliable informed consent

PRIOR CONCURRENT THERAPY:

* Previous treatment related toxicities should be resolved to grade 1 or better
* No other investigational agents within 14 days prior to the start of study
* No chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to start of study
* No major surgery within 2 weeks prior to start of study
* At least two weeks must have elapsed since the conclusion of radiation therapy and the start of gemcitabine hydrochloride, provided the acute effects of radiation treatment have been resolved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-01; Primary Completion 2010-08 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Advani, MD, Study Chair — The Cleveland Clinic
Locations (2):
- United States (2):
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were treated at the Cleveland Clinic or Duke University Medical Center during the years 2005-2008.
Pre-assignment Details: If </= 5 of the initial 18 patients enrolled achieved a CR, the study would be stopped. Accrual was not halted while follow-up of the first 18 evaluable patients was under way. Therefore, 24 patients were enrolled. Only 5 patients (21%) achieved a CR and therefore, the study was terminated.
Period: Overall Study
Arm/Group | Gemcitabine + Mitoxantrone
Started | 24
Completed | 23
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine + Mitoxantrone
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 51 [28 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Assumptions/ hypothesis: A Complete Response (CR) rate of 30% or less is unacceptable, and 50% or more is promising. A two-stage design will be used. Initially, 18 patients will be enrolled. If 5 or fewer achieve CR, the study will be stopped. Otherwise, an additional 22 patients will be accrued. Accrual was not halted while follow-up of the first 18 evaluable patients was under way. Therefore, 24 patients were enrolled. Four weeks is anticipated for observation for response. Only 5 patients (21%) achieved a CR and therefore, the study was terminated. Since response was assessed using the International Working Group criteria, a complete response was determined by Morphologic complete remission: A CR designation requires that the patient achieve the morphologic leukemia-free state and have an absolute neutrophil count of more than 1,000/μL and platelets of ≥ 100,000/μL, a cytogenic CR and a morphologic CR with incomplete blood count recovery (CRi).
Time Frame: 4 Weeks
Population: A total of 5 patients (21%) achieved a complete response.
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Mitoxantrone
Number analyzed (Participants) | 24
participants | 5

2. Secondary Outcome: Disease-free and Overall Survival
Time Frame: After a CR is achieved, patients are followed at 3 month intervals for disease progression and survival. If a patient has disease progression after achieving a CR, survival will be captured at 6 month intervals, typically for up to 5 years.
Population: 1 patient died on day 1 of protocol therapy (secondary to complications from AML).
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Mitoxantrone
Number analyzed (Participants) | 24
participants
  Patients dead >30 days post-tx, no relapse | 1
  Patients alive with no evidence of disease relapse | 4
  Patient death on Day 1 of Protocol Therapy | 1
  Patients dead >30 days post-tx, after relapse | 18

3. Secondary Outcome: Laboratory Correlates: Immunohistochemistry
Description: Percentage of patients who had a moderate-strong (2-3+) expression of multidrug resistance (MDR) genes by immunohistochemistry.
  * Multidrug resistance gene 1 (MDR1)
  * Equilibrative nucleoside transporter 2(SLC29A2)
Time Frame: Baseline
Population: 23 of 24 patients had available blocks for Immunohistochemical (IHC) analysis; Participants with the SLC29A2 Gene Expression (n=22)
Measure: Number; unit: percentage of participants
Arm/Group | Gemcitabine + Mitoxantrone
Number analyzed (Participants) | 23
percentage of participants
  Participants with GSTP1 Gene Expression | 70
  Participants with SLC29A2 Gene Expression | 55
  Participants with MRP1 Gene Expression | 43
  Participants with LRP1 Gene Expression | 35
  Participants with MDR1 Gene Expression | 22

4. Secondary Outcome: White Blood Cell Count at Time of Relapse
Time Frame: After a CR is achieved, patient will be followed at 3 month intervals for disease progression, typically for up to 5 years.
Measure: Median (Full Range); unit: cells per microliter
Arm/Group | Gemcitabine + Mitoxantrone
Number analyzed (Participants) | 24
cells per microliter | 3450 [800 to 233,500]

5. Primary Outcome: Duration of the First Complete Response
Time Frame: as for outcome 2
Population: Only 5 patients had a complete response, therefore on 5 patients were analyzed for this measure.
Measure: Median (Full Range); unit: months
Arm/Group | Gemcitabine + Mitoxantrone
Number analyzed (Participants) | 5
months | 7.3 [2.9 to 30.3]

6. Secondary Outcome: Percentage of Patients Making it to Bone Marrow Transplant.
Description: Assessing the number of patients who were able to have protocol treatment and have a bone marrow transplant after treatment.
Time Frame: After completion of protocol therapy
Measure: Number; unit: percentage of Patients completed a BMT
Arm/Group | Gemcitabine + Mitoxantrone
Number analyzed (Participants) | 24
percentage of Patients completed a BMT | 8

ADVERSE EVENTS:
Description: All Adverse Event (AE) / Serious Adverse Event (SAE) data grades were included together in data reporting; there was no differentiation between AEs and SAEs and no unexpected toxicities were seen. Since all grades were reported together, they are being listed as Serious for that reason.
Arm/Group | Gemcitabine + Mitoxantrone
Serious Adverse Events (participants affected / at risk) | 24/24
Other Adverse Events (participants affected / at risk) | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine + Mitoxantrone (N=24)
Fever or Infection (Infections and infestations) | 20
Rash (Skin and subcutaneous tissue disorders) | 19
Nausea (Gastrointestinal disorders) | 16
Pain (General disorders) | 16
Mucositis (Gastrointestinal disorders) | 14
Diarrhea (Gastrointestinal disorders) | 14
Fatigue (Musculoskeletal and connective tissue disorders) | 12
Abdominal Pain (Gastrointestinal disorders) | 9

LIMITATIONS AND CAVEATS:
If </= 5 of 1st 18 pts had a CR, study would stop (otherwise, another 22 pts would be accrued). Study would stop if >4 of 1st 10 or 10 of 1st 25 pts had unacceptable toxicity per protocol & Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No